CLINICAL TRIAL: NCT04288037
Title: Fetal Heart Rate Variability Compared to Doppler Flows in the Growth Restricted Fetus: a Cohort Study
Brief Title: Fetal Heart Rate Variability and Fetal Growth Restriction
Acronym: (FGR)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Snedkermester Sophus Jacobsen and hustru Astrid Jacobsens Foundation (Other); Hartmann Fonden (Other); Augustinus Fonden (Other); The Dagmar Marshall Foundation (Other); AP Moeller Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: fHRV_3
Record Dates: First submitted 2020-02-20; First posted 2020-02-27 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-02

CONDITIONS: Fetal Growth Retardation
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: fetal heart rate variability — observational study. no intervention

SUMMARY:
There is growing evidence in the field of fetal heart rate variability revealing the fetal neurological state. Furthermore, fetal heart rate variability has shown potential as fetal surveillance in fetal growth restriction.

This study aim to investigate the association between fetal heart rate variability and doppler flow changes in growth restricted fetuses.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnant women with estimated fetal weight below 2 standard deviations (2SD) of mean for gestational age corresponding to minus 22%. Fetal weight assessed by doppler ultrasound.

Exclusion Criteria:

* Fetal malformations

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women expecting a small for gestational age child. Danish.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Root mean square of successive inter beat interval differences RMSSD | 1/12-2020
  Time domain analysis
Standard deviation of normal to normal inter beat interval (SDNN) | 1/12-2020
  Time domain analysis
Low frequency power (LF-power) | 1/12-2020
  Spectral analysis
High frequency power (HF-power) | 1/12-2020
  Spectral analysis
Low frequency power/High frequency power (LF/HF) | 1/12-2020
  Spectral analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Arhus Universityhospital, Aarhus, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zizzo AR, Hansen J, Peteren OB, Molgaard H, Uldbjerg N, Kirkegaard I. Growth-restricted human fetuses have preserved respiratory sinus arrhythmia but reduced heart rate variability estimates of vagal activity during quiescence. Physiol Rep. 2022 Nov;10(22):e15458. doi: 10.14814/phy2.15458. PMID 36411966